CLINICAL TRIAL: NCT02778191
Title: Comparison of Concomitant Cisplatin Versus Carboplatin and 5-fluorouracil With Radiotherapy for Locally Advanced Head and Neck Squamous Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Collaborators: Amsterdam UMC, location VUmc (Other)
Responsible Party: Sponsor
Other Study IDs: 201501099
Record Dates: First submitted 2015-12-15; First posted 2016-05-19 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and neck squamous cell carcinoma; cisplatin; carboplatin; 5-fluorouracil
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Carboplatin; Fluorouracil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Concomitant cisplatin: Patients treated with concomitant cisplatin
  Interventions: Drug: cisplatin
- Carboplatin plus 5-FU: Patients treated with carboplatin plus 5-FU
  Interventions: Drug: carboplatin; Drug: 5-FU

INTERVENTIONS:
Drug: cisplatin — 100 mg/m2 day 1, 22 and 43
  Groups: Concomitant cisplatin
Drug: carboplatin — carboplatin 300-350 mg/m2 day 1, 22 and 43
  Groups: Carboplatin plus 5-FU
Drug: 5-FU — 5-FU 600 mg/m2 days 1-4, 22-25 and 43-46
  Groups: Carboplatin plus 5-FU

SUMMARY:
Concomitant chemoradiotherapy improves overall survival in patients with locally advanced head and neck squamous cell carcinoma (LA-HNSCC) compared to radiotherapy alone. Cisplatin 100 mg/m2 at day 1, 22 and 43 is widely used but results in considerable acute and late toxicity. Three cycles of carboplatin plus 5-fluorouracil (5-FU) is an accepted alternative but both chemotherapy regimens have not been compared prospectively. The aim of this study is to compare tolerability, efficacy, toxicity and quality of life in patients with LA-HNSCC treated with concomitant cisplatin and carboplatin plus 5-FU.

DETAILED DESCRIPTION:
This is a retrospective comparison of patients with LA-HNSCC treated with chemoradiotherapy at 2 tertiary care centers in the Netherlands (UMCG and VUmc), where one center routinely gives carboplatin plus 5FU (UMCG) and the other center (VUmc) uses high dose cisplatin as standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Stage III-IV LA-HNSCC of hypopharynx, oropharynx, larynx, oral cavity
* Primary treatment with concomitant chemoradiotherapy consisting of three-weekly cisplatin or carboplatin plus 5-FU
* Age ≤ 70 years
* No previous treatment for head and neck cancer
* No distant metastases

Exclusion Criteria:

* Previous treatment for head and neck cancer
* Distant metastases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced head and neck squamous cell carcinoma
Sampling Method: Probability Sample
Enrollment: 413 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Chemotherapy completion rate | 1 year
  The percentage of patients who completed 3 cycles of chemotherapy between both cohorts will be compared.

SECONDARY OUTCOMES:
Overall survival | 1 year
Progression free survival | 1 year
Distant metastases | 1 year
Grade 3-4 acute toxicity | 1 year
  retrospective data collection
Late toxicity | 1 year
  retrospective data collection
Quality of life | 1 year
  EORTC questionnaire QLQ C30
Quality of life | 1 year
  EORTC questionnaire HN35

CONTACTS AND LOCATIONS:
Overall Officials: S. Oosting, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - VUmc, Amsterdam
  - University Medical Center Groningen, Groningen